CLINICAL TRIAL: NCT05115903
Title: A Prospective, Randomized Biologic Tapering Study of TNF Inhibitors in Axial Spondyloarthritis
Brief Title: Biologic Tapering Study of TNF Inhibitors in Axial Spondyloarthritis
Acronym: BIOTAPE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Robert Inman, Principal Investigator, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-5211
Record Dates: First submitted 2021-10-28; First posted 2021-11-10 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Axial Spondyloarthritis
Keywords: spondyloarthritis; TNF inhibitors; tapering
MeSH Terms: conditions — Axial Spondyloarthritis; Spondylarthritis | interventions — Etanercept; Adalimumab; Certolizumab Pegol; golimumab; Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tapered doses of TNFi (Experimental): Tapering of TNFi through standardized increases in the dosing interval between drug administration. The tapering dose intervals for each TNFi are designed to decrease the dose from baseline by 75% for 12 weeks, 50% for 24 weeks, and 25% for 12 weeks
  Interventions: Drug: Tapered doses of TNFi
- Standard dose of TNFi (Active Comparator): Stable doses of TNFi according to the approved summary of product characteristics for biologic agents used in axial spondyloarthritis
  Interventions: Drug: Standard dose of TNFi

INTERVENTIONS:
Drug: Tapered doses of TNFi — To be given subcutaneously via a prefilled syringe/autoinjector (etanercept, adalimumab, certolizumab pegol, golimumab) or intravenously via infusion (infliximab) at increasing dose intervals as specified
  Other Names: etanercept 50 mg every 10 days (75% of baseline dose), 14 days (50%), 30 days (25%); adalimumab 40 mg every 3 weeks (75%), 4 weeks (50%), 16 weeks (25%); certolizumab pegol 200 mg 3 weeks (75%), 4 weeks (50%), 16 weeks (25%); golimumab 50 mg every 6 weeks (75%), 8 weeks (50%), 16 weeks (25%); infliximab 5 mg/kg every 8 weeks (75%), 12 weeks (50%), 16 weeks (25%)
  Arms: Tapered doses of TNFi
Drug: Standard dose of TNFi — To be given subcutaneously via a prefilled syringe/autoinjector (etanercept, adalimumab, certolizumab pegol, golimumab) or intravenously via infusion (infliximab)
  Other Names: etanercept 50 mg every 7 days; adalimumab 40 mg every 2 weeks; certolizumab pegol 200 mg every 2 weeks; golimumab 50 mg every 4 weeks; infliximab 5 mg/kg every 6 weeks
  Arms: Standard dose of TNFi

SUMMARY:
Current evidence on tapering of tumor necrosis factor inhibitors (TNFi) in axial spondyloarthritis (axSpA) is still hampered by heterogeneity in tapering regimens, selection and performance biases, and lack of data on optimized treatment dosing strategies especially in real-world clinical settings. This study aims to contribute to the ongoing investigation of disease-activity-guided tapering of TNFi in axSpA in the form of a prospective, randomized controlled trial.

DETAILED DESCRIPTION:
This is a 48-week randomized, controlled, open-label, non-inferiority trial of patients with radiographic or non-radiographic axial spondyloarthritis. The study will include 156 patients with inactive disease or low disease activity (LDA) for at least 6 months on a TNFi at the time of randomization.

Participants will be randomized using a 1:1 ratio to either the tapered-dose arm or the standard-dose arm of TNFi. Progressive tapering of TNFi according to a predefined protocol will be allowed as long as the patient is able to maintain inactive disease or LDA during the study period. We hypothesize that, in patients with 6 months or more of inactive or low-activity axial spondyloarthritis, tapered-dose TNFi are non-inferior to standard-dose TNFi in sustaining the disease state for at least 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Adult axSpA patients satisfying the 2009 Assessment of SpondyloArthritis International Society (ASAS) Classification Criteria
* Currently enrolled in the SPARCC Program with successful completion of standard data collection protocol in the Spondylitis Clinic of UHN-Toronto Western Hospital
* Have sustained inactive disease or LDA with an ASDAS of <2.1 or BASDAI <4 for at least 6 months
* On a stable dose of a TNFi (infliximab, etanercept, adalimumab, certolizumab pegol, or golimumab)
* Must not be pregnant

Exclusion Criteria:

* Adults axSpA patients with active extra-articular manifestations such as inflammatory bowel disease, psoriasis, and/or uveitis
* Have comorbidities that may preclude clinical assessment (i.e. fibromyalgia or other chronic pain syndromes; chronic inflammatory diseases other than axSpA)
* Have diagnosed psychiatric or personality disorders
* Pregnant
* Not enrolled in the Spondyloarthritis Research Consortium of Canada (SPARCC) Program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients able to maintain inactive disease or low disease activity, defined as Ankylosing Spondylitis Disease Activity Score (ASDAS) <1.3 to 2.1 or Bath Ankylosing Spondylitis Disease Activity Score (BASDAI) of <4 on tapered-dose TNFi | Weeks 12, 24, 36, and 48
  The ASDAS and BASDAI are measures of axial spondyloarthritis disease activity for the past week. The ASDAS has 5 components scored from 0 to 10 (none to very severe). The following formula is used to compute for the ASDAS: (0.121 × back pain score) +(0.058 × score for duration of morning stiffness) + (0.11 × patient global assessment score) + (0.073 × peripheral pain/swelling score) + (0.579 × log(CRP+1)). The scores range from 0 (no disease activity) to infinity (being determined by the level of CRP). The disease is considered inactive if the final score is <1.3, and low if <2.1.
  The BASDAI consists of six items, with each item being scored from 0 ("none") to 10 ("very severe"). The final BASDAI scores ranges from 0 to 10, with lower scores indicating lower disease activity. A BASDAI of <4 indicates inactive or low disease.
  As opposed to ASDAS, BASDAI does not include CRP in its formula. Either ASDAS or BASDAI is acceptable in clinical practice.

SECONDARY OUTCOMES:
Proportion of patients experiencing a disease flare by ASDAS or BASDAI | Up to Week 48
  Flare is defined in this study as either of the following:
  1. loss of inactive disease or LDA (ASDAS ≥2.1 or BASDAI ≥4) - see definitions above
  2. minimal clinically important worsening, defined as an increase in ASDAS by ≥0.9 on two consecutive visits
Proportion of patients with functional limitation measured using the Bath Ankylosing Spondylitis Functional Index (BASFI) | Up to Week 48
  The BASFI measures the degree of functional limitation. It is composed of a set of 10 questions relating to activities during the past week. Each item is scored from 0 ("easy") to 10 ("impossible"). The final BASFI is the mean of the 10 scores with the total score ranging from 0 to 10. Lower scores indicate better physical function.
Mean quality of life in the tapered-dose arm vs. the standard-dose arm measured using the Ankylosing Spondylitis Quality of Life (ASQoL) questionnaire | Up to Week 48
  The ASQoL measures health-related quality of life (HRQoL) in subjects with axial spondyloarthritis. The final ASQoL score ranges from 0 to 18, with higher scores indicating worse HRQoL.
Proportion of patients with impaired work productivity and activity measured using the Work Productivity and Activity Impairment Questionnaire for Ankylosing Spondylitis (WPAI:SpA) questionnaire | Up to Week 48
  The WPAI:SpA consists of 6 questions to determine employment status, hours missed from work because of SpA, hours missed from work for other reasons, hours actually worked, the effect of SpA on work productivity while at work, and the effect of SpA on activities outside of work. The 4 scores derived include percentage of absenteeism, percentage of presenteeism (reduced productivity while at work), an overall work impairment combining absenteeism and presenteeism, and percentage of impairment in activities performed outside of work. The computed percentage for each sub-scale ranges from 0 to 100. Higher scores indicate greater impairment and less productivity.
Proportion of patients with radiographic progression, defined as an increase in the modified Stoke Ankylosing Spondylitis Spine Score (mSASSS) by 2 units | Baseline and Week 48
  The mSASSS measures the sum of the lumbar and cervical spine score from 0 (no change) to 72 (progression). The score is derived from grading of the anterior aspect of the vertebral bodies of the lumbar spine (T12 to S1) and the cervical spine (C2 to T1). Grading is as follows: 0 (normal), 1 (erosion, sclerosis, or squaring), 2 (syndesmophyte), 3 (bridging syndesmophyte), or N (vertebral body not evaluable).
Proportion of patients needing concomitant medication | Up to Week 48
  Concomitant medications will include NSAIDs, conventional synthetic DMARDs, and/or targeted synthetic DMARDs used during the study period
Proportion of patients with any related severe adverse event | Up to Week 48
  Severe adverse event, defined as serious infections requiring systemic antibiotic use and/or hospitalization assessed to be at least possibly related to TNFi use or withdrawal
Factors predicting flare | Up to Week 48
  Factors including but not be limited to the following: sex, human leukocyte antigen (HLA)-B27 status, disease duration, duration of remission, ASDAS at the start of taper, and MRI findings at the time of taper

CONTACTS AND LOCATIONS:
Overall Officials: Robert D. Inman, MD, Principal Investigator — University Health Network - Toronto Western Hospital
Locations (1):
- University Health Network - Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Braun J, Brandt J, Listing J, Zink A, Alten R, Golder W, Gromnica-Ihle E, Kellner H, Krause A, Schneider M, Sorensen H, Zeidler H, Thriene W, Sieper J. Treatment of active ankylosing spondylitis with infliximab: a randomised controlled multicentre trial. Lancet. 2002 Apr 6;359(9313):1187-93. doi: 10.1016/s0140-6736(02)08215-6. PMID 11955536
- [Background] van der Heijde D, Kivitz A, Schiff MH, Sieper J, Dijkmans BA, Braun J, Dougados M, Reveille JD, Wong RL, Kupper H, Davis JC Jr; ATLAS Study Group. Efficacy and safety of adalimumab in patients with ankylosing spondylitis: results of a multicenter, randomized, double-blind, placebo-controlled trial. Arthritis Rheum. 2006 Jul;54(7):2136-46. doi: 10.1002/art.21913. PMID 16802350
- [Background] Inman RD, Davis JC Jr, Heijde Dv, Diekman L, Sieper J, Kim SI, Mack M, Han J, Visvanathan S, Xu Z, Hsu B, Beutler A, Braun J. Efficacy and safety of golimumab in patients with ankylosing spondylitis: results of a randomized, double-blind, placebo-controlled, phase III trial. Arthritis Rheum. 2008 Nov;58(11):3402-12. doi: 10.1002/art.23969. PMID 18975305
- [Background] Navarro-Compan V, Plasencia-Rodriguez C, de Miguel E, Balsa A, Martin-Mola E, Seoane-Mato D, Canete JD. Anti-TNF discontinuation and tapering strategies in patients with axial spondyloarthritis: a systematic literature review. Rheumatology (Oxford). 2016 Jul;55(7):1188-94. doi: 10.1093/rheumatology/kew033. Epub 2016 Mar 21. PMID 26998860
- [Background] Gratacos J, Pontes C, Juanola X, Sanz J, Torres F, Avendano C, Vallano A, Calvo G, de Miguel E, Sanmarti R; REDES-TNF investigators. Non-inferiority of dose reduction versus standard dosing of TNF-inhibitors in axial spondyloarthritis. Arthritis Res Ther. 2019 Jan 8;21(1):11. doi: 10.1186/s13075-018-1772-z. PMID 30621746
- [Background] Zhang T, Zhu J, He D, Chen X, Wang H, Zhang Y, Xue Q, Liu W, Xiang G, Li Y, Yu Z, Wu H. Disease activity guided stepwise tapering or discontinuation of rhTNFR:Fc, an etanercept biosimilar, in patients with ankylosing spondylitis: a prospective, randomized, open-label, multicentric study. Ther Adv Musculoskelet Dis. 2020 Jun 2;12:1759720X20929441. doi: 10.1177/1759720X20929441. eCollection 2020. PMID 32536984
- [Background] Lawson DO, Eraso M, Mbuagbaw L, Joanes M, Aves T, Leenus A, Omar A, Inman RD. Tumor Necrosis Factor Inhibitor Dose Reduction for Axial Spondyloarthritis: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Arthritis Care Res (Hoboken). 2021 Jun;73(6):861-872. doi: 10.1002/acr.24184. PMID 32166872